CLINICAL TRIAL: NCT05832593
Title: Immunohistochemical Expression of Excision Repair Cross Complementation Group 1 (ERCC1) in Laryngeal Squamous Cell Carcinoma and Its Correlation With Response to Radiotherapy.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Mohamed Abdel hameed, Adminstrator in Pathology department, Faculty Of Medicine, Assiut University
Other Study IDs: ERCC1 in laryngeal cancers
Record Dates: First submitted 2023-04-15; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Laryngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Other: Immunohistochemistry
- Group 2
  Interventions: Other: Immunohistochemistry

INTERVENTIONS:
Other: Immunohistochemistry — Immunohistochemical expression of ERCC1

SUMMARY:
1. Determine the correlation between immunohistochemical expression of ERCC1 in laryngeal cancer cells with clinico-pathological variables.
2. Assess the correlation between ERCC1 expression and response to radiotherapy.

DETAILED DESCRIPTION:
The global burden of laryngeal cancer increased during the past 3 decades. A total number of 210,606 new cases of laryngeal cancer have been diagnosed in 2017 (2.76 new cases per 100,000 inhabitants) worldwide, with a prevalence of 1.09 million cases (14.33 cases per 100,000 inhabitants), accounting for as many as 126,471 deaths (1.66 per 100,000 inhabitants). The incidence and prevalence have both increased by 12.0% and 23.8%, respectively during the past 3 decades, whilst mortality has declined by approximately 5 %.

In Egypt, laryngeal cancer represents 5.7% of all body malignancies and 38.7% of the head and neck malignancies.

Squamous cell carcinoma is the most common histologic variant and accounts for 85-95% of all malignant tumors of the larynx. According to World Health Organization it is the second most common malignancy of the upper aerodigestive tract. It occurs more in people above 40 years of age and more common in males.

The larger number of laryngeal cancer cases originate from the glottic region (i.e., approximately two-third), followed by the supraglottic area (about 30%), whilst trans-glottic and purely subglottic tumors are generally less frequent.

Excision repair cross-complementation group 1 (ERCC1) is a key DNA repair gene in the nucleotide excision repair pathway which is activated in the repair of intra- and interstrand DNA crosslink.

Ionizing radiation (IR) acts directly or indirectly to cause various forms of deoxyribonucleic acid (DNA) damage in cells. DNA damage repair is initiated after the cell is genetically damaged. Nucleotide-excision repair (NER) is one of the ways of DNA repair. ERCC1 is a structure-specific endonuclease that cut DNA at single-stranded/double-stranded junctions with a specific polarity.

There is some clinical evidence suggesting that ERCC1 status (ERCC1 mRNA expression, ERCC1 protein expression, and ERCC1 polymorphisms) is associated with platinum-based therapy efficacy in some kinds of cancers.

In a previous meta-analysis, ERCC1 protein low expression status detected by immunohistochemical methods significantly correlated with higher response to platinum-based chemotherapy in ovarian cancers.

Another meta-analysis evaluated non-small cell lung cancer patients treated with platinum-based chemoradiation showed that both low tumoral mRNA and protein levels were associated with a better response rate and overall patient survival.

In head and neck squamous cell carcinomas, the available studies have a conflict in results. Of six studies evaluating the relation between ERCC1 status and outcomes of head and neck cancer patients, three showed positive and another three were with negative results.

ELIGIBILITY:
Inclusion Criteria:

* Stage: All stages of laryngeal squamous cell carcinoma.
* Grade: Both high and low grades.
* Patients treated with radiotherapy.
* Normal laryngeal tissue as a control.

Exclusion Criteria:

* • Patients with deficient clinical data.

  * Patients treated with chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with laryngeal squamous cell carcinoma that will be treated with radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Investigate the immunohistochemical expression of ERCC1 in laryngeal squamous cell carcinoma and correlate between its expression and response to radiotherapy. | 12 months
  Immunohistochemical staining for ERCC1 using monoclonal antibodies on paraffin blocks with immunoperoxidase technique will be assessed to detect expression of ERCC1 in laryngeal squamous cell carcinoma. Evaluation of ERCC1 expression depends on evaluating intensity and extent of staining.

REFERENCES:
- [Background] Nocini R, Molteni G, Mattiuzzi C, Lippi G. Updates on larynx cancer epidemiology. Chin J Cancer Res. 2020 Feb;32(1):18-25. doi: 10.21147/j.issn.1000-9604.2020.01.03. PMID 32194301
- [Background] Fasunla AJ, Ogundoyin OA, Onakoya PA, Nwaorgu OG. Malignant tumors of the larynx: Clinicopathologic profile and implication for late disease presentation. Niger Med J. 2016 Sep-Oct;57(5):280-285. doi: 10.4103/0300-1652.190596. PMID 27833247
- [Background] Hoffman HT, Porter K, Karnell LH, Cooper JS, Weber RS, Langer CJ, Ang KK, Gay G, Stewart A, Robinson RA. Laryngeal cancer in the United States: changes in demographics, patterns of care, and survival. Laryngoscope. 2006 Sep;116(9 Pt 2 Suppl 111):1-13. doi: 10.1097/01.mlg.0000236095.97947.26. PMID 16946667
- [Background] Markou K, Christoforidou A, Karasmanis I, Tsiropoulos G, Triaridis S, Constantinidis I, Vital V, Nikolaou A. Laryngeal cancer: epidemiological data from Nuorthern Greece and review of the literature. Hippokratia. 2013 Oct;17(4):313-8. PMID 25031508
- [Background] Avinash Tejasvi ML, Maragathavalli G, Putcha UK, Ramakrishna M, Vijayaraghavan R, Anulekha Avinash CK. Impact of ERCC1 gene polymorphisms on response to cisplatin based therapy in oral squamous cell carcinoma (OSCC) patients. Indian J Pathol Microbiol. 2020 Oct-Dec;63(4):538-543. doi: 10.4103/IJPM.IJPM_964_19. PMID 33154302
- [Background] Jiang C, Guo Y, Li Y, Kang J, Sun X, Wu H, Feng J, Xu Y. The association between the ERCC1/2 polymorphisms and radiotherapy efficacy in 87 patients with non-small cell lung cancer. J Thorac Dis. 2021 May;13(5):3126-3136. doi: 10.21037/jtd-21-755. PMID 34164203
- [Background] Vilmar A, Sorensen JB. Excision repair cross-complementation group 1 (ERCC1) in platinum-based treatment of non-small cell lung cancer with special emphasis on carboplatin: a review of current literature. Lung Cancer. 2009 May;64(2):131-9. doi: 10.1016/j.lungcan.2008.08.006. Epub 2008 Sep 19. PMID 18804893
- [Background] Bohanes P, Labonte MJ, Lenz HJ. A review of excision repair cross-complementation group 1 in colorectal cancer. Clin Colorectal Cancer. 2011 Sep;10(3):157-64. doi: 10.1016/j.clcc.2011.03.024. Epub 2011 Apr 28. PMID 21855036
- [Background] Langer CJ. Exploring biomarkers in head and neck cancer. Cancer. 2012 Aug 15;118(16):3882-92. doi: 10.1002/cncr.26718. Epub 2012 Jan 26. PMID 22281752
- [Background] Li FY, Ren XB, Xie XY, Zhang J. Meta-analysis of excision repair cross-complementation group 1 (ERCC1) association with response to platinum- based chemotherapy in ovarian cancer. Asian Pac J Cancer Prev. 2013;14(12):7203-6. doi: 10.7314/apjcp.2013.14.12.7203. PMID 24460276
- [Background] Chen S, Zhang J, Wang R, Luo X, Chen H. The platinum-based treatments for advanced non-small cell lung cancer, is low/negative ERCC1 expression better than high/positive ERCC1 expression? A meta-analysis. Lung Cancer. 2010 Oct;70(1):63-70. doi: 10.1016/j.lungcan.2010.05.010. Epub 2010 Jun 11. PMID 20541281
- [Background] Jun HJ, Ahn MJ, Kim HS, Yi SY, Han J, Lee SK, Ahn YC, Jeong HS, Son YI, Baek JH, Park K. ERCC1 expression as a predictive marker of squamous cell carcinoma of the head and neck treated with cisplatin-based concurrent chemoradiation. Br J Cancer. 2008 Jul 8;99(1):167-72. doi: 10.1038/sj.bjc.6604464. PMID 18594541
- [Background] Fountzilas G, Bamias A, Kalogera-Fountzila A, Karayannopoulou G, Bobos M, Athanassiou E, Kalogeras KT, Tolis C, Tsekeris P, Papakostas P, Vamvouka C, Zaramboukas T, Kosmidis P, Zamboglou N, Misailidou D. Induction chemotherapy with docetaxel and cisplatin followed by concomitant chemoradiotherapy in patients with inoperable non-nasopharyngeal carcinoma of the head and neck. Anticancer Res. 2009 Feb;29(2):529-38. PMID 19331199
- [Background] Handra-Luca A, Hernandez J, Mountzios G, Taranchon E, Lacau-St-Guily J, Soria JC, Fouret P. Excision repair cross complementation group 1 immunohistochemical expression predicts objective response and cancer-specific survival in patients treated by Cisplatin-based induction chemotherapy for locally advanced head and neck squamous cell carcinoma. Clin Cancer Res. 2007 Jul 1;13(13):3855-9. doi: 10.1158/1078-0432.CCR-07-0252. PMID 17606717
- [Background] Fountzilas G, Kalogera-Fountzila A, Lambaki S, Wirtz RM, Nikolaou A, Karayannopoulou G, Bobos M, Kotoula V, Murray S, Lambropoulos A, Aravantinos G, Markou K, Athanassiou E, Misailidou D, Kalogeras KT, Skarlos D. MMP9 but Not EGFR, MET, ERCC1, P16, and P-53 Is Associated with Response to Concomitant Radiotherapy, Cetuximab, and Weekly Cisplatin in Patients with Locally Advanced Head and Neck Cancer. J Oncol. 2009;2009:305908. doi: 10.1155/2009/305908. Epub 2009 Dec 29. PMID 20066159
- [Background] Koh Y, Kim TM, Jeon YK, Kwon TK, Hah JH, Lee SH, Kim DW, Wu HG, Rhee CS, Sung MW, Kim CW, Kim KH, Heo DS. Class III beta-tubulin, but not ERCC1, is a strong predictive and prognostic marker in locally advanced head and neck squamous cell carcinoma. Ann Oncol. 2009 Aug;20(8):1414-9. doi: 10.1093/annonc/mdp002. Epub 2009 May 25. PMID 19468031
- [Background] Hayes M, Lan C, Yan J, Xie Y, Gray T, Amirkhan RH, Dowell JE. ERCC1 expression and outcomes in head and neck cancer treated with concurrent cisplatin and radiation. Anticancer Res. 2011 Dec;31(12):4135-9. PMID 22199271